CLINICAL TRIAL: NCT03249909
Title: A Clinical Investigation to Study the Effect of Exufiber Ag+ and Other Gelling Fibre Dressings on Wound Exudate and Bioburden in Medium to High Exuding Wounds
Brief Title: Evaluation of Exufiber Ag+ and Other Gelling Fibre Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exufiber Ag+ 01
Record Dates: First submitted 2017-08-06; First posted 2017-08-15 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2019-03

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Subjects were to be assigned in the following order:
  * Eligible Subjects 1 to 50 were to be assigned to the Exufiber Ag+ cohort
  * Eligible Subjects 51 to 65 were to be assigned to Exufiber
  * Eligible Subjects 66 to 85 were to be assigned to Aquacel Ag Extra
  * Eligible Subjects 86 to 105 were to be assigned to Exufiber Ag+ on eligible pressure ulcer subjects
  The statistical analysis of the groups treated will be analysed separately with the same statistical methods.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Exufiber Ag + (Other): Gelling fibre dressing with silver to treat chronic wounds, acute wounds, and pressure ulcers. Data from these groups were analyzed separately with no comparative analysis.
  Interventions: Device: Exufiber Ag+; Device: Exufiber; Device: Aquacel Ag Extra
- Exufiber (Other): Gelling fibre dressing without silver to treat chronic wounds, acute wounds, and pressure ulcers. Data from these groups were analyzed separately with no comparative analysis.
  Interventions: Device: Exufiber Ag+; Device: Exufiber; Device: Aquacel Ag Extra
- Aquacel® Ag Extra (Other): Gelling fibre dressing with silver to treat chronic wounds, acute wounds, and pressure ulcers. Data from these groups were analyzed separately with no comparative analysis.
  Interventions: Device: Exufiber Ag+; Device: Exufiber; Device: Aquacel Ag Extra

INTERVENTIONS:
Device: Exufiber Ag+ — gelling fibre dressing with silver
Device: Exufiber — gelling fibre without silver
Device: Aquacel Ag Extra — gelling fibre with silver

SUMMARY:
Investigate impact of gelling fiber dressings on handling exudate in medium to high exuding wounds

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Both gender ≥ 18 years old
* From Medium to High exuding wound

Exclusion Criteria:

* Known allergy or hypersensitivity to any of the treatment dressings
* Pregnant or lactating females
* Subjects with a target wound that is ≤1 cm2
* Subjects with a target wound that is a full thickness burn
* Subjects with a target wound that is a full thickness pressure ulcer
* Subjects with known immunodeficiency
* Subject taking systemic antibiotics for wound infection
* Subject were the target wound is located on an infected limb interfered by minimal blood flow in the opinion of the investigator
* Subject with a target wound with unexplored enteric fistula
* Subjects who in the opinion of the investigator, will have problems following the protocol
* Subjects needing treatment with oxidizing agents such as hypochlorite solutions or hydrogen peroxide
* Previously enrolled in the present investigation
* Inclusion in other ongoing investigations at present that would preclude the subject from participating in this investigation as judged by the investigator
* Involvement in the planning and conduct of the clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, MAS, Principal Investigator — University of Miami
Locations (8):
- United States (8):
  - Midwestern University, Glendale, Arizona
  - Center for Clinical Research, Inc., San Francisco, California
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Boise VA Medical Center (Boise VAMC) M, Boise, Idaho
  - Northwell Health, Lake Success, New York
  - Jobst Vascular Institue (JVI), Toledo, Ohio
  - Serena Group Research Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total enrolment was 109 subjects from 9 sites in the US, and was completed between 11 AUG 2017 and 12 JUN 2019.
Pre-assignment Details: All enrolled subjects were assigned to a treatment group and treated in compliance with the Instructions For Use. No subject was excluded from the intent-to-treat (ITT) and safety population during analysis.
Groups:
- Exufiber Ag+; Aquacel Ag Extra: Gelling fiber dressing with silver to treat 'chronic wounds', 'acute wounds', and 'pressure ulcers' for the purpose of data analysis. Data from these groups were analyzed separately with no comparative analysis.
- Exufiber: Gelling fiber dressing without silver to treat 'chronic wounds', 'acute wounds', and 'pressure ulcers' for the purpose of data analysis. Data from these groups were analyzed separately with no comparative analysis.
Period: Overall Study
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Started | 78 | 15 | 16
Completed | 72 | 14 | 16
Not Completed | 6 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exufiber Ag+: Exufiber Ag+ included treatment for 'chronic wounds', 'acute wounds', and 'pressure ulcers' for the purpose of data analysis. Data from these groups were analyzed separately with no comparative analysis.
- Exufiber: Exufiber included treatment for 'chronic wounds' and 'acute wounds' for the purpose of data analysis. Data from these groups were analyzed separately with no comparative analysis.
- Aquacel Ag Extra: Aquacel Ag Extra included treatment for 'chronic wounds' and 'acute wounds' for the purpose of data analysis. Data from these groups were analyzed separately with no comparative analysis.
- Total: Total of all reporting groups
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra | Total
Number analyzed (Participants) | 78 | 15 | 16 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.9) | 56.9 (16.8) | 56.6 (11.5) | 61.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 9 | 4 | 42
  Male | 49 | 6 | 12 | 67
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 78 | 15 | 16 | 109
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (8.8) | 35.8 (11.2) | 35.8 (10.9) | 33.7 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Exudate Status From Baseline to Last Visit
Description: The primary endpoint measures exudate status based on dressing condition in categorical variables: Dry, Moist, Wet, Saturated, Leaking. Analysis of the change in exudate status (Decrease, Equal/Unchanged, Increase) from baseline to 4 weeks in the treatment groups was performed with a two-sided Sign test on the Intent To Treat (ITT) population at significance level 0.05.
  If a subject had missing values at 4 weeks (Visit 5), last observation carried forward (LOCF) was applied from Visit 2 (1 week). Three subjects treated with Exufiber Ag+ did not have evaluable data: 2 of the subjects did not complete a Visit 2 (1 week) or later visits (both subjects with a chronic wound); 1 subject (with a chronic wound) only completed the investigation until Visit 2, however no exudate status data were reported at Visit 2 for that subject. One subject treated with Exufiber did complete a Visit 2 (1 week) or later visit.
Time Frame: 4 weeks (28 days) or earlier if the wound is dry or healed
Population: Intent To Treat (ITT) population with evaluable data to analyze change from baseline to last visit (n=75 for Exufiber Ag+; n=14 for Exufiber; n=16 for Aquacel Ag Extra)
Measure: Count of Participants; unit: Participants
Arm/Group | Exufiber Ag + | Exufiber | Aquacel® Ag Extra
Number analyzed (Participants) | 75 | 14 | 16
Participants
  Decreased exudate status | 27 | 3 | 7
  Unchanged exudate status | 40 | 6 | 8
  Increased exudate status | 8 | 5 | 1
Statistical Analysis 1: Comparison: Exufiber Ag +; Test type: Non-Inferiority — Analysis of the change in exudate status (Decrease, Equal/Unchanged, Increase) from baseline to 4 weeks in the treatment groups with the two-sided Sign test on the Intent To Treat (ITT) population at 95% confidence interval; p = 0.0019, Sign test

2. Secondary Outcome: 4-Week Wound Status
Description: The overall wound status was evaluated by the Nurse/Investigator in ordered, categorical variables (Stagnated, Aggravated, Same as baseline, Improved, Healed), and presented with number of participants at week 4 (28 days).
  The total number (n) represents the total number of subjects included at the study visit; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat population with available data for this data point at Visit 5, or 4 weeks (28 days), is n=60 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: At 4 weeks (28 days)
Population: Intent to Treat population with available data at 4 weeks (28 days) (n=60 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra)
Measure: Count of Participants; unit: Participants
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 60 | 13 | 12
Participants
  Stagnated | 2 | 1 | 1
  Aggravated | 5 | 3 | 0
  Sames as baseline | 1 | 1 | 3
  Improved | 48 | 7 | 6
  Healed | 4 | 1 | 2

3. Secondary Outcome: Wound Area Reduction (mm^2)
Description: Wound area was calculated as an ellipse, i.e. Area = (Longest length/2) x (Longest width/2) x π, and was measured by a third-party validated software system. To account for subjects requiring debridement, wound area presented here are pooled data for wounds not debrided and after debridement.
  The total number (n) represents the total number of subjects included at the study visit with evaluable data; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing). Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), or earlier if the wound is dry or healed, is n=59 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: Total treatment period of 4 weeks (28 days) or earlier if the wound is dry or healed
Population: Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), or earlier if the wound is dry or healed, is n=59 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 59 | 13 | 12
mm^2 | -388.4 (707.6) | -296.3 (2567.7) | -274.7 (546.1)

4. Secondary Outcome: Frequency of Dressing Changes Between Visits
Description: Frequency of dressing change was evaluated by the Nurse/Investigator. Dressing changes for each dressing were to be performed at least weekly, in line with the IFU and schedule of assessment.
  Values over 1 indicate dressing changes were required between study follow up visits, for any reason.
Time Frame: Total treatment period of 4 weeks (28 days) or earlier if the wound is dry or healed
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: dressing changes / 7 days
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 78 | 15 | 16
dressing changes / 7 days | 1.36 (1.77) | 0.511 (0.633) | 3.56 (1.56)

5. Secondary Outcome: Tissue Type of Wound Bed
Description: Measurement of tissue types were collected separately, including necrotic tissue, sloughy tissue, granulation tissue, and epithelialized tissue. The change in percent of tissue type from baseline to 4 weeks are presented with number and percentages.
  The total number (n) represents the total number of subjects included at the study visit with evaluable data; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), or earlier if the wound is dry or healed, is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: Total treatment period of 4 weeks (28 days) or earlier if the wound is dry or healed
Population: Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), or earlier if the wound is dry or healed, is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Measure: Mean (Standard Deviation); unit: change in percentage
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 61 | 13 | 12
change in percentage
  Change in percent of necrotic tissue | 2.13 (14.73) | 1.54 (23.04) | 2.5 (8.66)
  Change in percent of sloughy tissue | -6.48 (28.20) | -2.69 (40.08) | -0.833 (6.686)
  Change in percent of granulation tissue | -5.33 (37.14) | -12.7 (40.1) | -18.3 (39.7)
  Change in percent of epithelialisation | 11.4 (29.2) | 13.8 (29.6) | 16.7 (38.9)

6. Secondary Outcome: Status of the Wound and Peri-wound Skin From Baseline to Last Visit: Malodour
Description: Malodour was evaluated by the Nurse/Investigator in ordered categorical variables, None, Slight, Moderate, Strong. The Sign test was used for analysis of reported changes within groups from baseline to 4 weeks (Decrease, Equal/Unchanged, Increase), and described with number and percentages of reported changes.
  The total number (n) represents the total number of subjects included at the study visit; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat (ITT) population with available data to analyze change from baseline to Visit 5, at 4 weeks (28 days), is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: Total treatment period of 4 weeks (28 days)
Population: Intent to Treat (ITT) population with available data to analyze change from baseline to Visit 5, at 4 weeks (28 days), is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Measure: Count of Participants; unit: Participants
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 61 | 13 | 12
Participants
  Decrease | 3 | 0 | 0
  Equal/Unchanged | 45 | 8 | 9
  Increase | 13 | 5 | 3

7. Secondary Outcome: Status of the Wound and Peri-wound Skin From Baseline to Last Visit: Redness/Irritation
Description: Redness/Irritation under and outside the Primary dressing was evaluated by the Nurse/Investigator in and recorded as present (Yes) or not present (No). The Sign test was used for analysis of reported changes within groups from baseline to 4 weeks (Decrease, Equal/Unchanged, Increase), and presented with number and percentages of reported changes.
  The total number (n) represents the total number of subjects included at the study visit; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat (ITT) population with available data to analyze change from baseline to Visit 5, at 4 weeks (28 days), is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: Total treatment period of 4 weeks (28 days)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 61 | 13 | 12
Participants
  Decrease | 8 | 0 | 1
  Equal/Unchanged | 53 | 13 | 9
  Increase | 0 | 0 | 2

8. Secondary Outcome: Status of the Wound and Peri-wound Skin From Baseline to Last Visit: Maceration
Description: Maceration under and outside the Primary dressing was evaluated by the Nurse/Investigator in and recorded as present (Yes) or not present (No). The Sign test was used for analysis of reported changes within groups from baseline to 4 weeks (Decrease, Equal/Unchanged, Increase), and presented with number and percentages of reported changes.
  The total number (n) represents the total number of subjects included at the study visit; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat (ITT) population with available data to analyze change from baseline to Visit 5, at 4 weeks (28 days), is n=61 for Exufiber Ag+; n=13 for Exufiber; n=12 for Aquacel Ag Extra.
Time Frame: Total treatment period of 4 weeks (28 days)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 61 | 13 | 12
Participants
  Decrease | 16 | 0 | 5
  Equal/Unchanged | 39 | 13 | 7
  Increase | 6 | 0 | 0

9. Secondary Outcome: Handling and Technical Performance of the Dressing
Description: Handling and technical performance of the dressings were evaluated by the Nurse/Investigator in ordered categorical variables, Very Poor, Poor, Good, Very Good, and NA. We have presented the percentage of study participants reported with the category variable, Very Good, for each question at 4 weeks (28 days).
  The total number (n) represents the total number of subjects included at the study visit with evaluable data; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), is n=63 for Exufiber Ag+; n=15 for Exufiber; n=16 for Aquacel Ag Extra.
Time Frame: At 4 weeks (28 days)
Population: Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), is n=63 for Exufiber Ag+; n=15 for Exufiber; n=16 for Aquacel Ag Extra.
Measure: Number; unit: % of subjects
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 63 | 15 | 16
% of subjects
  Ease of application of dressing | 57.8 | 100.0 | 66.7
  Ease of removal of dressing without moistening | 56.4 | 85.7 | 63.6
  Removal in one piece | 64.3 | 92.9 | 63.6
  Ability to absorb exudate | 55.4 | 92.9 | 55.6
  Ability to absorb blood | 59.2 | 92.9 | 55.6
  Ability to retain exudate | 60.7 | 92.9 | 55.6
  Ability to retain slough | 55.6 | 92.9 | 55.6
  Ability to clean wound bed | 49.2 | 92.9 | 44.4
  Ability to retain balanced moist environment | 50.0 | 92.9 | 55.6
  Conformability to wound | 48.3 | 92.9 | 60.0
  Overall experience | 51.7 | 92.9 | 60.0

10. Secondary Outcome: Comfort, Conformability, and Acceptability of the Dressings by Subject
Description: Comfort, conformability, and acceptability of the dressings were evaluated by the Subject Participant in ordered categorical variables, Very Poor, Poor, Good, Very Good, and NA. We have presented the percentage of study participants reported with the category variable, Very Good, for each question at 4 weeks (28 days) or earlier if the wound dried or healed.
  The total number (n) represents the total number of subjects included at the study visit with evaluable data; data were not always recorded for every subject, at every visit, for every data parameter (i.e. some data/answers are missing); Intent to Treat population with available data at Visit 5, or 4 weeks (28 days), is n=63 for Exufiber Ag+; n=15 for Exufiber; n=16 for Aquacel Ag Extra.
Time Frame: At 4 weeks (28 days) or earlier if the wound is dry or healed
Population: as for outcome 9
Measure: Number; unit: % of subjects
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
Number analyzed (Participants) | 63 | 15 | 16
% of subjects
  Comfort while wearing | 44.3 | 57.1 | 66.7
  Ease of mobility | 41.0 | 64.3 | 66.7
  Primary dressing remained in place | 49.2 | 64.3 | 58.3
  No stinging or burning | 87.5 | 85.7 | 100.0
  Overall experience | 45.6 | 64.3 | 63.6

ADVERSE EVENTS:
Time Frame: All adverse event data were collected for a period of 2 years, throughout enrollment and follow-up of this study
Description: There were no reports of death in any group throughout the study, and no reports of SAEs in the Exufiber group.
Arm/Group | Exufiber Ag+ | Exufiber | Aquacel Ag Extra
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 7/78 | 0/15 | 1/16
Other Adverse Events (participants affected / at risk) | 14/78 | 5/15 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exufiber Ag+ (N=78) | Exufiber (N=15) | Aquacel Ag Extra (N=16)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization following syncopal episode
Arteriovenous fistula (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for right arm fistula
Revisional transmetatarsal amputation right foot (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for transmetatarsal amputation on right foot with full thickness wound along surgical site.
Infection on non-study foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — In-patient hospitalization for infection on non-study foot
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for pneumonia
Kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for kidney injury
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for shortness of breath
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for cellulitis of the lower limb
Inability to eat (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — In-patient hospitalization for inability to eat
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exufiber Ag+ (N=78) | Exufiber (N=15) | Aquacel Ag Extra (N=16)
Cellulitis of non-study wound (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cellulitis of study wound (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cold (General disorders) | 1 (1) | 0 (0) | 0 (0) — Cold, or flu-like symptoms
Exacerbation of congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infection of the study wound (Infections and infestations) | 2 (2) | 1 (2) | 1 (1)
Itching of the non-study wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Maceration in study wound (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
New ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in study wound (General disorders) | 4 (4) | 0 (0) | 0 (0)
Pain not related to study wound (General disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This clinical investigation was limited in that it was non-comparative and based on a limited number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03249909/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03249909/ICF_001.pdf